CLINICAL TRIAL: NCT07177976
Title: Comparative Effects of Pilates Breathing and Pursed Lip Breathing on Chest Expension and Peak Expiratory Flow Rate in Patients With Chronic Obstructive Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/91
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive (COPD)
Keywords: Chest expansion; peak expiratory flow rate; dyspnea
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group (interventional group) wil receive Pilates breathing along with pharmacological management and the other group (control group) will perform Pursed-lip breathing along with pharmacological management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients in this group will receive Pilates breathing techniques along with pharmacological management for total of 3 weeks.
  Two sessions per week will be supervised by physiotherapist and 5 days at home. A home diary will be provided in order to ensure and follow-up of the participants are performing breathing exercises at home.
  Interventions: Procedure: Pilates Breathing Technique along with standard pharmacological management
- Group B (Experimental): Patients in this group will receive Pursed-lip breathing along with pharmacological management for 3 weeks.
  Two sessions per weeek will be supervised by physiotherapist and 5 days at home.
  A home diary will be provided in order to ensure and follow-up of the participants that they are performing breathing exercises at home.
  Interventions: Procedure: Pursed-lip breathing along with pharmacological management

INTERVENTIONS:
Procedure: Pilates Breathing Technique along with standard pharmacological management — Patients in this group will receive pilates breathing technique along with pharmacological management.
  A total 3 weeks protocol will be followed in which 2 seesions per week will be supervised by physiotherapist and 5 days at home.
  Pilates breathing will be performed in sitting or supine position. The patient will place a hand over the Lower Posterior rib Cage and inhale through the nose.
  While breathing they will actively contract the Transverse Abdominis (TrA) as if preparing for punch or holding in urine and engaging the pelvic floor muscles.
  Arms: Group A
Procedure: Pursed-lip breathing along with pharmacological management — Patient in this group will receive pursed-lip breathing along with pharmacological management. A total 3 weeks protocol will be followed in which 2 sessions per week will be supervised by physiotherapist and 5 days at home.
  The patient will sit comfortably with straight back and relaxed shoulders. They will inhale slowly through the nose, with a deep relaxed breath, and then exhale slowly through the pursed lips, as if blowing out a candle. The exhalation should take 2-3 times longer than inhalation. This breathing cycle will be repeated with a focus on slow and relaxed breathing.
  Pharmacological management: Patient will receive medications as per prescribed by pulmonologist
  Arms: Group B

SUMMARY:
Chronic Obstructive Pulmonary Disease is a particular type of irreversible disease that may damage or obstruct airways and make it difficult to breath. This respiratiry condition may lead to shallow breathing.

Breathing exercisers help to manage hyperventilation often seen in COPD patients. To handle respiratory complications patients are advised to practice breathing techniques along with pharmacological management

DETAILED DESCRIPTION:
Chronic Obstructive pulmonary Disease is a particular type of irreversible disease that may damage or obstruct airways and make it difficult to breath. This respiratory condition may lead to shallow breathing.

Breathing exercises help to manage hyperventilation often seen in copd patients. To handle respiratory complications patients are advised to practice brathing techniques along with pharmacological management.

Total 46 participants are allocated divided into two group. Group A will perform Pilates breathing along with pharmacological management and group B will perform Pursed-lip breathing along with pharmacological management.

Hence objective of study is to compare the effects of pilates breathing techniques along with pharmacological management versus pursed-lip breathing along with pharmacological management on chest expansion, peak expiratory flow rate, dyspnea and quality of life in patients with chronic obstructive lung disease

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-64 years
* Both genders (male and female)
* Grade 1-3 on mMRC scale of dyspnea
* COPD mild stage according to global initiative for chronic obstructive lung disease (GOLD) classification; Mild = FEV1 greater than or equal to 80% predicted

Exclusion Criteria:

* Moderate, severe and very severe stage of COPD according to GOLD classification
* Patients having acute exerbation of COPD
* Patients diagnosed with acute infection
* Patients unable to follow command and instructions

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Chest Expansion | 03 weeks
  Evaluation will be done using inch tape (inches) for Chest Expansion
Peak expiratory flow rate | 03 weeks
  Evaluation will be done by using Peak flow meter
Dyspnea | 03 weeks
  Evaluation will be done by using Modified Medical Research Council Dyspnea Scale (mMRC)

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, 44000, Rawalpindi, Pakistan